CLINICAL TRIAL: NCT05413135
Title: A Phase 2 Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of ARO-APOC3 in Adults With Dyslipidemia
Brief Title: Study of ARO-APOC3 in Adults With Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AROAPOC3-2003
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARO-APOC3 (Experimental): 1 dose of ARO-APOC3 by subcutaneous (sc) injection every 3 months
  Interventions: Drug: ARO-APOC3

INTERVENTIONS:
Drug: ARO-APOC3 — ARO-APOC3 Injection

SUMMARY:
This is an open-label extension of the parent studies AROAPOC3-2001 and AROAPOC3-2002. Adult participants with dyslipidemia who completed the blinded 12-month period from either parent study and continued to meet eligibility criteria had the option to be enrolled into this study. Eligible enrolled participants initially received open-label ARO-APOC3 every three or six months at the assigned dose level of the parent study until a final dose of 25 mg was selected, at which point all participants transitioned to the selected dosing regimen of 25 mg every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are nonpregnant, nonlactating and do not plan to become pregnant during the study
* Able and willing to provide written informed consent
* Completed the 48-week study treatment period in the parent study

Exclusion Criteria:

* Subject was permanently discontinued from ARO-APOC3 in the parent study due to elevated glycated hemoglobin (HbA1c), aspartate aminotransferase (AST) or alanine aminotransferase (ALT)
* Any new condition or worsening of existing condition or any other situation that would make the subject unsuitable for enrollment, could interfere with the subject participating in or completing the study, would make it difficult to comply with protocol requirements or put the subject at additional safety risk
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Through 24 months

SECONDARY OUTCOMES:
Change from Baseline in Fasting Triglycerides (TG) Over Time | Through 24 months
Percent Change from Baseline in Fasting TG Over Time | Through 24 months
Change from Baseline in Apolipoprotein (Apo) C-III Over Time | Through 24 months
Percent Change from Baseline in ApoC-III Over Time | Through 24 months
Change from Baseline in Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) Over Time | Through 24 months
Percent Change from Baseline in Fasting Non-HDL-C Over Time | Through 24 months
Change from Baseline in Fasting High-Density Lipoprotein-Cholesterol (HDL-C) Over Time | Through 24 months
Percent Change from Baseline in Fasting HDL-C Over Time | Through 24 months
Change from Baseline in Fasting Total Apolipoprotein B (ApoB) Over Time | Through 24 months
Percent Change from Baseline in Fasting Total ApoB Over Time | Through 24 months
Change from Baseline in Fasting Low-Density Lipoprotein-Cholesterol (LDL-C) Over Time Using Ultracentrifugation | Through 24 months
Percent Change from Baseline in Fasting LDL-C Over Time Using Ultracentrifugation | Through 24 months

CONTACTS AND LOCATIONS:
Locations (60):
- United States (30):
  - Clinical Research Site 1, Beverly Hills, California
  - Clinical Research Site 2, Northridge, California
  - Clinical Research Site 3, Palm Springs, California
  - Clincal Research Site 4, Boca Raton, Florida
  - Clinical Research Site 5, Fort Lauderdale, Florida
  - Clinical Research Site 8, Miami, Florida
  - Clinical Research Site 6, Miami, Florida
  - Clinical Research Site 9, Miami Springs, Florida
  - Clinical Research Site 10, Pembroke Pines, Florida
  - Clinical Research Site 11, Port Orange, Florida
  - Clinical Research Site 12, Dunwoody, Georgia
  - Clinical Research Site 13, Minneapolis, Minnesota
  - Clinical Research Site 14, Tupelo, Mississippi
  - Clinical Research Site 15, Omaha, Nebraska
  - Clinical Research Site 16, Las Vegas, Nevada
  - Clinical Research Site 17, Long Island City, New York
  - Clinical Research Site 18, New Windsor, New York
  - Clinical Research Site 19, New York, New York
  - Clinical Research Site 20, Morehead City, North Carolina
  - Clinical Research Site 21, Fargo, North Dakota
  - Clinical Research Site 22, Marion, Ohio
  - Clinical Research Site 23, Maumee, Ohio
  - Clinical Research Site 24, Oklahoma City, Oklahoma
  - Clinical Research Site 25, Greenville, South Carolina
  - Clinical Research Site 26, Chattanooga, Tennessee
  - Clinical Research Site 29, Houston, Texas
  - Clinical Research Site 27, Houston, Texas
  - Clinical Research Site 28, Houston, Texas
  - Clinical Research Site 30, San Antonio, Texas
  - Clinical Research Site 31, Manassas, Virginia
- Australia (7):
  - Clinical Research Site 32, Camperdown, New South Wales
  - Clinical Research Site 33, Milton, Queensland
  - Clinical Research Site 34, Sippy Downs, Queensland
  - Clinical Research Site 35, Adelaide, South Australia
  - Clinical Research Site 36, Clayton, Victoria
  - Clinical Research Site 37, Joondalup, Washington
  - Clinical Research Site 38, Nedlands, Washington
- Canada (5):
  - Clinical Research Site 39, Concord, Ontario
  - Clinical Research Site 40, London, Ontario
  - Clinical Research Site 41, Chicoutimi, Quebec
  - Clinical Research Site 43, Montreal, Quebec
  - Clinical Research Site 44, Québec, Quebec
- Hungary (6):
  - Clinical Research Site 46, Balatonfüred
  - Clinical Research Site 47, Békéscsaba
  - Clinical Research Site 48, Debrecen
  - Clinical Research Site 49, Gyöngyös
  - Clinical Research Site 50, Komárom
  - Clinical Research Site 51, Nyíregyháza
- Netherlands (3):
  - Clinical Research Site 53, Amsterdam
  - Clinical Research Site 54, Sneek
  - Clinical Research Site 55, Zwijndrecht
- New Zealand (3):
  - Clinical Research Site 58, Papatoetoe, Aukland
  - Clinical Research Site 56, Christchurch
  - Clinical Research Site 57, Christchurch
- Poland (6):
  - Clinical Research Site 59, Bydgoszcz
  - Clinical Research Site 64, Lodz
  - Clinical Research Site 63, Lodz
  - Clinical Research Site 60, Oświęcim
  - Clinical Research Site 61, Poznan
  - Clinical Research Site 62, Rzeszów

IPD SHARING:
Plan to Share IPD: No